CLINICAL TRIAL: NCT00469898
Title: A Phase II Trial of Carboplatin and Irinotecan (CPT-11) as First-Line Therapy for Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Irinotecan and Carboplatin as First-Line Therapy in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leora Horn, MD, Assistant Professor of Medicine; Assistant Director, Educator Development Program; Clinical Director, Thoracic Oncology Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC THO 0321; VU-VICC-THO-0321
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2011-03-23 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental): Lung cancer patients will be treated for four 3-week cycles (12 weeks) in the absence of progressive disease, unacceptable toxicity, or withdrawal of patient consent. Up to two additional cycles may be administered at the discretion of the treating physician. If at treatment withdrawal the disease has responded or is stable, the patient will continue to be followed for efficacy (i.e. until progressive disease)at 8 week intervals. Following the diagnosis of progressive disease, patients will be followed every two months for survival.
  Interventions: Drug: Carboplatin; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: Carboplatin — Carboplatin dosage calculation to be given on day 1, every 21 days:
  Carboplatin (mg) = (AUC of 5) x (GFR + 25)
  *up to 6 cycles at physician's discretion
  Other Names: Paraplatin
Drug: irinotecan hydrochloride — 50 mg/m2 IV on days 1 and 8 every 21 days
  Should be infused IV over 30- 90 minutes.
  Other Names: Irinotecan; Camptosar; CPT-11

SUMMARY:
RATIONALE: The general results of combining irinotecan and platin-based chemotherapies have been very encouraging. As the toxicity profile associated with carboplatin is preferable over cisplatin it is our expectation that patients and physicians would prefer to use this combination if it is equally or more efficacious. To date there has been no agreement regarding the optimal combination of these agents. Based on the trials described in the protocol and our experience with carboplatin/irinotecan in the treatment of non-small cell lung cancer the present trial will utilize a 21-day cycle of irinotecan 50 mg/m2 given on days 1 and 8 and carboplatin AUC 5 (based on the Calvert formula) on day 1.

PURPOSE: This phase II trial is studying how well giving irinotecan together with carboplatin works as first-line therapy in treating patients with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To examine the anti-tumor efficacy of the combination of Irinotecan (CPT-11) and Carboplatin as first-line therapy as assessed by response rate in patients with chemo-naïve extensive stage small cell lung cancer.

Secondary

* Determine the safety, tolerability, and feasibility of this regimen in these patients.
* Determine the time to progression in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter, open-label study.

Patients receive irinotecan IV over 30-90 minutes on days 1 and 8 and carboplatin IV on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 54 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer (SCLC)

  * Extensive stage small cell lung cancer
* Must have ≥ 1 unidimensionally measurable lesion (longest diameter to be recorded) ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan

  * Lesion cannot be from a previously irradiated area
  * Lesions that are considered nonmeasurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
    * Tumor lesions in a previously irradiated area
* No brain metastasis or carcinomatous meningitis unless stable and asymptomatic

PATIENT CHARACTERISTICS

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* ANC ≥ 1,500/mm³
* Platelet count > 100,000/mm³
* Serum bilirubin ≤ 1.5 mg/dL
* AST/SGOT ≤ 2.5 times upper limit of normal (ULN) (or ≤ 5 times ULN if liver metastases present)
* Serum creatinine ≤ 2.0 mg/dl
* Hemoglobin ≥ 9.0 g/dl

Exclusion Criteria:

* CNS metastasis excluded unless: stable and asymptomatic
* Coexisting medical condition that would preclude study compliance
* Patients with Gilbert's disease
* Uncontrolled diabetes mellitus, defined as random blood sugar ≥ 300 mg/dl or > 16.6 mmol/L
* Patients who do not discontinue phenytoin, phenobarbitol, carbamazipine, or other enzyme-inducing anticonvulsant drugs at least 7 days prior to first treatment dose on study. Gabapentin is permitted
* Patients who do not discontinue St. John's Wort prior to first treatment dose on study.
* Patients who are pregnant or breast feeding
* Concomitant second active malignancy except for any in situ cancer or adequately treated basal cell or squamous cell skin cancer or any cancer from which the patients has been disease-free for at least 2 years
* No administration of any prior systemic anticancer therapy for extensive stage SCLC such as: chemotherapy, antibody therapy, immunotherapy, gene therapy, vaccine therapy, cytokine therapy, or other experimental agents. Concurrent use of other anticancer therapy including inhibitors of vascular endothelial or epidermal growth factor pathways is prohibited. Prior radiation is allowed
* Symptomatic brain metastasis or carcinomatous meningitis

PRIOR CONCURRENT THERAPY:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-12; Primary Completion 2008-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horn, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (8):
- United States (7):
  - Owensboro Medical Health System, Owensboro, Kentucky
  - Memorial Health Care System, Chattanooga, Tennessee
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - St. Thomas Health Services, Nashville, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
- British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period = 2/18/2004 through 1/23/2007
Pre-assignment Details: A total of 54 people signed consent to take part in the study. Of those, 3 were found to be ineligible and 1 withdrew before beginning the study.
Period: Overall Study
Arm/Group | Therapeutic Intervention
Started | 50
Completed | 25
Not Completed | 25
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 4
Not completed — Death | 4
Not completed — Disease progression | 9
Not completed — Decreased performance status | 1

BASELINE CHARACTERISTICS:
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 59.5 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 45
  Canada | 5

OUTCOME MEASURES:

1. Primary Outcome: Patient Response
Description: Patient response to treatment:
  Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started Complete response (CR): disappearance of all target lesions Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD
Time Frame: 1.66 months (average duration, on treatment date to best response date)
Measure: Number; unit: participants
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 50
participants
  Complete Response | 2
  Not Assessed | 1
  Not Evaluable | 2
  Partial Response | 27
  Progressive Disease | 12
  Stable Disease | 1
  Unknown | 5

2. Secondary Outcome: Number of Patients With Adverse Events
Description: Number of participants with adverse events, according to grade of event, using the NCI Common Toxicity Criteria (version 2.0) grading system to assign a grade to each event
Time Frame: date off treatment or progression of disease, up to 18 weeks
Measure: Number; unit: participants
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 50
participants
  Grade 1 | 13
  Grade 2 | 26
  Grade 3 | 29
  Grade 4 | 10
  Grade 5 | 4

3. Secondary Outcome: Time to Progression
Description: Time to progression in months
Time Frame: 9.9 months (on study date to progression)
Population: Patients who has progression
Measure: Median (Full Range); unit: Months
Units Other Than Participants: Non censoring patients
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 50
Number analyzed (Non censoring patients) | 40
Months | 5 [1 to 17]

4. Secondary Outcome: Overall Survival
Time Frame: On study date to death
Measure: Median (Full Range); unit: Months
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 50
Months | 9 [0 to 42]

ADVERSE EVENTS:
Arm/Group | Therapeutic Intervention
Serious Adverse Events (participants affected / at risk) | 26/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Intervention (N=50)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Arthritis pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Asystole/Possible PE (Cardiac disorders) | 1 (1)
Back and shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac infarction (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Death due to disease progression (General disorders) | 2 (2)
Death, unknown cause (General disorders) | 1 (1)
Decrease in platelet count (Investigations) | 5 (5)
Decreased neutrophil count (Investigations) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Fainting (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased hemoglobin (Investigations) | 4 (4)
Left proximal humerus fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8)
Peri-rectal abscess (Gastrointestinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post-obstructive pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Weight loss (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes